CLINICAL TRIAL: NCT04903704
Title: Pulmonary HypERtenSion and Measurement of Exercise caPacIty REmotely: the PERSPIRE Study
Brief Title: Pulmonary Hypertension and Measurement of Exercise Capacity Remotely
Acronym: PERSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH21477
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sit to Stand testing (Other): Participants will undergo an ISWT in the hospital setting. This test is a standard of clinical care and it is essential to the patient assessment on their clinical visit. This test will therefore be conducted first in all cases.
  They will be allowed a 30 minute rest before undertaking the 1MSTS test.
  Clinical observations (heart rate, blood pressure, oxygen saturations) will be taken before and after both tests. Heart rate and oxygen saturations will be monitored during both tests.
  Patient reported measures of dyspnoea and perceived exertion will be recorded on completion of both tests.
  Adverse events e.g. dizziness, syncope or the participant becoming unwell be recorded.
  Descriptive and inferential statistical analysis will be used to determine the safety of 1MSTS in the hospital setting and comparability between 1MSTS and ISWT for participants. We will also examine comparability between 1MSTS outcomes and other available routinely collected clinical data.
  Interventions: Diagnostic Test: 1 Minute Sit to Stand Test

INTERVENTIONS:
Diagnostic Test: 1 Minute Sit to Stand Test — Participants are asked to stand repeatedly from a chair for one minute without the use of their arms for support. The number of completed repetitions is counted.

SUMMARY:
Background

Hospital-based walking exercise tests are routinely used in patients with pulmonary hypertension to assess functional ability and disease progression over time. We are seeing a greater emphasis on non-face-to-face clinical assessments, where such tests cannot be conducted. It is important to identify alternative tests which can be which can be conducted by patients at home and used to support clinical decision making.

Aim

To test the safety of the 1-minute sit-to-stand test in patients with pulmonary hypertension and its comparability with hospital-based walking exercise tests.

Methods

A sample of 75 patients attending hospital appointments will carry out an Incremental Shuttle Walk Test, followed by a 1-minute sit-to-stand test after a 30 minute rest. Data will be analysed for safety and comparability between the 2 tests.

In the event of favourable findings (safety and comparability) from the hospital-based testing, a further sample of patients will be asked to perform the 1-minute sit-to-stand test in the home setting

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a progressive condition affecting the circulation to the lungs from the heart. It is a rare condition and Sheffield Pulmonary Vascular Diseases Unit (SPVDU) is the largest of 7 adult specialist pulmonary hypertension centres, caring for 1900 patients, or 30% of the pulmonary hypertension patients treated in the UK. Measures of how well patients tolerate exercise and their functional abilities are widely established in pulmonary hypertension. This includes hospital-based assessments such as Incremental Shuttle Walk Test (ISWT - a "beep" test which requires patients to walk progressively faster until they cannot continue) and 6 minute walking test (how far patients can walk in 6 minutes), which are included in international risk guidelines for PH. At SPVDU patients attend clinic appointments at intervals ranging from 3 -12 months; an ISWT is conducted at every clinic visit and the results are used to monitor functional progress over time.

This study will seek to establish the safety of the 1-minute sit-to-stand test and its comparability to the Incremental Shuttle Walk Test. Participants will be recruited as part of their standard clinic visit to SPVDU. They will undergo their standard clinical Incremental Shuttle Walk Test. This test is a standard of clinical care and its essential to the patient assessment on their clinical visit and will therefore be conducted first in all cases. They will be allowed a 30 minute rest before undertaking the 1-minute sit-to-stand test.

It is standard at SPVDU that patients undertake the Incremental Shuttle Walk Test without supplemental oxygen - standardised protocols allow for this if repeat tests follow the same procedure. Patients are advised that they should stop the activity when they feel they can no longer continue. The same protocol will be adopted for the 1-minute sit-to-stand test.

Clinical observations (heart rate, blood pressure, oxygen saturations) will be taken before and after both tests. Heart rate and oxygen saturations will be monitored during both tests. Patient reported measures of breathlessness and perceived exertion will be recorded on completion of both tests.

Adverse events e.g. dizziness, syncope or the participant becoming unwell be recorded. Adverse event data will be monitored and analysed to determine the safety of the 1MSTS test. To assist in the planning or potential next stages of the study, participants will be asked if they have access to equipment that would support home monitoring e.g. tape measure, BP monitor, pulse oximeter, weighing scales, video calling.

Data collected during the testing will be analysed, along with other routinely collected clinical data to determine the comparability of the 1MSTS test with with ISWT and other clinical features.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH)

Exclusion Criteria:

* mobility significantly impaired by musculoskeletal or neurological co-morbidities; learning difficulties or cognitive impairment that would prohibit informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Sit to stand repititions | Counted during testing
  The number of completed sit to stand repetitions in 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Carol Keen, Principal Investigator — Physiotherapist
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No